CLINICAL TRIAL: NCT02829463
Title: Magnetic Resonance Imaging of Infrapatellar Fat Pad in Osteoarthritis and Controls
Brief Title: MRI of Infrapatellar Fat Pad in Osteoarthritis
Acronym: IPFP-MRI
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: JY201507
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- osteoarthritis patients: 3.0 Tesla Magnetic resonance imaging was analyzed. It's the documentation from the outpatients and inpatients with osteoarthritis. It's not the intervention the study applied, but the subjects' disease demands.
  Interventions: Radiation: Magnetic resonance imaging
- healthy controls: 3.0 Tesla Magnetic resonance imaging was analyzed. It's the documentation from the outpatients and inpatients without osteoarthritis. It's not the intervention the study applied, but the subjects' non-osteoarthritis knee symptom demands.
  Interventions: Radiation: Magnetic resonance imaging

INTERVENTIONS:
Radiation: Magnetic resonance imaging — 3.0 T Magnetic resonance imaging of knee joints. It does not harm the subjects.

SUMMARY:
In this study, the investigators use the clinical documentation and imaging data of MRI to do research. Clinical subjects were divided into two groups: osteoarthritis patients and healthy controls without osteoarthritis. Differences of MRI data were studied between two groups.

DETAILED DESCRIPTION:
In this study, the investigators applied high precision MRI technique (with as less as a slice thickness of 0.35 mm and without inter-slice gap), and calculated not only the IPFP maximal sagittal area and IPFP volume, but also the quantitated signal, and compared the differences between healthy controls and osteoarthritis patients. This is an observational cross-sectional study without specific interventions to the subjects. MRI is a regular examination in our hospital. And all subjects are included for the reasons of osteoarthritis (need MRI) and healthy controls (pain but not osteoarthritis, also need MRI). The investigator does not assign specific interventions to the subjects of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical knee osteoarthritis;
* The healthy controls who require MRI test.

Exclusion Criteria:

* Contraindications to magnetic resonance imaging;
* Rheumatoid arthritis patients;
* Gout;
* Hemophilic arthritis;
* Subjects who take non-steroidal anti-inflammatory drugs (NSAIDs);
* Subjects who take lipid-lowering agents;
* Subjects who have the history of knee trauma;
* Subjects who have the history of knee operation;
* Subjects who have the disease of musculoskeletal tumor near knee;
* Subjects who have joint loose bodies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who come to see doctors requiring knee MRI test.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinshen He, MD, Principal Investigator — Department of Orthopaedic Surgery, Third Xiangya Hospital of Central South University
Locations (1):
- Jinshen He, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pan F, Han W, Wang X, Liu Z, Jin X, Antony B, Cicuttini F, Jones G, Ding C. A longitudinal study of the association between infrapatellar fat pad maximal area and changes in knee symptoms and structure in older adults. Ann Rheum Dis. 2015 Oct;74(10):1818-24. doi: 10.1136/annrheumdis-2013-205108. Epub 2014 May 15. PMID 24833783
- [Background] Han W, Aitken D, Zhu Z, Halliday A, Wang X, Antony B, Cicuttini F, Jones G, Ding C. Signal intensity alteration in the infrapatellar fat pad at baseline for the prediction of knee symptoms and structure in older adults: a cohort study. Ann Rheum Dis. 2016 Oct;75(10):1783-8. doi: 10.1136/annrheumdis-2015-208360. Epub 2015 Nov 26. PMID 26612337

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Osteoarthritis Patients | Healthy Controls
Started | 59 | 62
Completed | 59 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osteoarthritis Patients | Healthy Controls | Total
Number analyzed (Participants) | 59 | 62 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.2) | 38.8 (13.6) | 49.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 23 | 33 | 56
BMI [Median (Standard Deviation); unit: kg/(m^2)] | 24.7 (3.5) | 22.6 (4.4) | 23.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Infrapatellar Fat Pad Volume in MRI
Time Frame: collect the data within 24 hours after the subjects did the MRI
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Osteoarthritis Patients | Healthy Controls
Number analyzed (Participants) | 59 | 62
mm^3 | 25154.96 (4865.37) | 29202.39 (7242.63)

ADVERSE EVENTS:
Arm/Group | Osteoarthritis Patients | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/62
Other Adverse Events (participants affected / at risk) | 0/59 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes